CLINICAL TRIAL: NCT01731262
Title: Preliminary Study of Sonic Hedgehog Signaling Pathway in the Pathogenesis of Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Shangling Zhu, Post-Graduate, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 中大附三医伦[2012]2-75号
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Arthritis, Rheumatoid; Neovascularization, Pathologic; Synovitis
Keywords: Arthritis, Rheumatoid; Sonic hedgehog protein, human; Neovascularization, Pathologic; Synovitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Neovascularization, Pathologic; Synovitis

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RA group: expression of Shh pathway associated factors from peripheral blood mononuclear cells or synovial tissues will be detected
- control group: expression of Shh pathway associated factors from peripheral blood mononuclear cells or synovial tissues will be detected

SUMMARY:
Rheumatoid arthritis(RA) with a high incidence and high morbidity, the pathogenesis has not been fully elucidated. Fibroblast-like synovial cells excessive proliferation and synovial angiogenesis is the most important cause of RA synovitis and joint destruction. Our study was to find the role of Sonic Hedgehog(SHH) pathway in regulating proliferation of fibroblast-like synovial cells and modulating excess angiogenesis of synovial tissue.

DETAILED DESCRIPTION:
4ml blood from active RA patients(n=35) and healthy volunteers (n=35) will be collected

* peripheral blood mononuclear cells will be detached
* messenger ribonucleic acid expression of Sonic Hedgehog pathway associated factors in both groups will be detected

Synovial tissues from 4 RA patients and 4 patients with traumatic or meniscal injury who need to carry out knee joint replacement operation will be collected

* inflammatory feature of synovial tissue will be observed
* the expression of Shh, Ptch1, Gli1 and Smo in synovial tissue will be detected by immunohistochemistry assay
* fibroblast-like synoviocytes will be cultured from synovial tissue of RA patients

ELIGIBILITY:
Inclusion Criteria:

* definitely diagnosed
* the disease is active (DAS28>3.2)

Exclusion Criteria:

* combined with severe organ dysfunction
* combined with other rheumatic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents of south China
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
mRNA expression | 1 day (December 15, 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Jianlin Huang, PhD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University